CLINICAL TRIAL: NCT01228630
Title: Randomized Clinical Study for Efficacy Assessment Between Cloratadd-D, Loratadine + Pseudoephedrine (Coated Pill), Produced by EMS S/A Laboratories and Allegra-D , Produced by Sanofi-Aventis for Patients With Perennial Allergic Rhinitis.
Brief Title: Effectiveness of Two Preparations of Loratadine + Pseudoephedrine in Patients With Perennial Allergic Rhinitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: EMS S/A (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOREMS0810
Record Dates: First submitted 2010-10-18; First posted 2010-10-26 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Perennial Allergic Rhinitis
Keywords: rhinitis, loratadine, coated pill
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis | interventions — Loratadine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cloratadd-D (Experimental): Loratadine 5 mg + 120 mg of sulfate pseudoephedrina and coated tablet of placebo (identical to comparator drug). The patients receive one pill of treatment every 12 hours ( to get up and going to bed), of a glass of water.
  Interventions: Drug: Cloratadd-D
- Allegra-D (Active Comparator): Loratadine 5 mg + 120 mg of sulfate pseudoephedrina and coated tablet of placebo (identical to test drug). The patients receive one pill of treatment every 12 hours ( to get up and going to bed), of a glass of water.
  Interventions: Drug: Allegra-D

INTERVENTIONS:
Drug: Cloratadd-D — The patients receive one pill of treatment every 12 hours ( to get up and going to bed), of a glass of water.
  Other Names: Loratadine + pseudoephedrine
  Arms: Cloratadd-D
Drug: Allegra-D — The patients receive one pill of treatment every 12 hours ( to get up and going to bed), of a glass of water.
  Other Names: Loratadine + pseudoephedrine
  Arms: Allegra-D

SUMMARY:
The loratadine-pseudoephedrine combination has proven to be more effective than the use of these individual components. This prospective, randomized, double-blind and paralel study, in which patients with perennial allergic rhinitis receive one of loratadine + pseudoephedrine association drug for treatment of signs and symptoms during 4 weeks.

DETAILED DESCRIPTION:
The effectiveness of treatment in each drug group will be evaluate by global improvement of signs (nasal mucous edema, ocular hyperemia, nasal secretion) and symptoms (itching eye, tearing,itching nose, itching on the palate) of perennial allergic rhinitis, after 4 weeks of treatment. Symptoms as rhinorrhea, nasal congestion, itching nose, sneezing and itching eye were considered as secondary efficacy endpoint, along with the questionnaire of quality of life SF-36. Safety evaluation data will include report of all adverse events (including type, frequency, instensity, seriousness, severity and action taken related to investigational product) reported by patients, parents or legal responsible, ou observed by Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Comply with all the purposes and procedures of the study by signing and dating the IC own free will. In the case of minors, the document should be signed and dated by the parent or legal guardian;
* Have age over 12 years, regardless of gender, ethnicity or social class;
* Present clinical status of perennial allergic rhinitis from mild to moderate;
* Present clinical status with at least 12 months of evolution;
* Submit the examination of IgE elevation (above 100KU / L).

Exclusion Criteria:

* Have participated in any experimental study or have taken any experimental drug in the 12 months preceding the start of the study;
* Pregnant or lactating women;
* Have made use of:

  1. Intranasal or systemic corticosteroids in the month before inclusion;
  2. Intranasal cromolyn in the two weeks preceding inclusion;
  3. Intranasal or systemic decongestants in the 03 days preceding inclusion;
  4. Intranasal antihistamines or systemic in the 03 days preceding the survey;
  5. Loratadine in the 10 days preceding the survey.
* have any disease or anatomical abnormality in the upper airways which could jeopardize the analysis of data, for example, tumors or severe septal deviations;
* History of smoking in the 03 months preceding the inclusion;
* History of alcohol or illicit drugs;
* History of liver disease or kidney disease;
* Electric current asthma or gift last year;
* Table of uncontrolled hypertension;
* Patients with heart disease or who use drugs for the cardiovascular system that is suffering interference of the drugs studied, for example, β-blockers;
* Patients with flu-like symptoms or fever of unknown origin, defined current or within last 07 days;
* Clinical diagnosis of rhinitis is not that kind of allergic and perennial;
* Be patient with sensitivity to loratadine, pseudoephedrine sulfate, or any components of the formula;
* Estimated travel or displacement of the southeast for more than 50% of monitoring.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms evaluated by a PHYSICIAN | 28 days of treatment.
  Signs of swelling of nasal mucosa,ocular hyperemia and nasal discharge. Symptoms of itchy eyes, watery eyes,itchy nose and itching of the palate. These signs and symptoms will be assessed during 04 scheduled visits: -7 days, 0 day, 7 days and 28 days.

SECONDARY OUTCOMES:
Symptoms reported by PATIENTS | 28 days of treatment.
  Symptoms of runny nose,nasal congestion, itchy nose, sneezing, quality of life.These signs and symptoms will be assessed during 04 scheduled visits: -7 days, 0 day, 7 days and 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Tikara Shimizu, PI, Principal Investigator — LAL Clinica Pesquisa e Desenvolvimento Ltda
Locations (1):
- Lal Clínica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It believed that after the data analysis and presentation to the IRC, all data will become public.